CLINICAL TRIAL: NCT04583137
Title: Buffered vs Plain Lidocaine for Local Nasal Anesthesia
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kfir Siag (Other)
Responsible Party: Sponsor-Investigator, Kfir Siag, Dr, Kfir Siag; Principal Investigator; Department of Otolaryngology-Head and neck surgery, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EMC-20-0185
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia, Local
Keywords: Nasal Sprays, Lidocaine, Bicarbonate, Local anesthesia

STUDY DESIGN:
Intervention Model Description: trial containing two groups. The first group receives an intranasal solution of lidocaine combined with bicarbonate. The second group receives intranasal plain lidocaine. After a measured time of 5 minutes, all patients will attend a TFL examination. The patients will fill the first questionnaire immediately after the procedure, a second questionnaire by telephone after one hour, and the third questionnaire by telephone after a one-month follow-up.
  Sample size was calculated using data from a previous publication of local soft tissue injection with buffered lidocaine5. This estimation power analysis showed that for VAS average and standard deviation were 3.5±1.4 for the lidocaine group and 2.5±1.4 for the second group given lidocaine with bicarbonate. In order to achieve a statistical power of 90% and significance of p<0.05 a sample of 40 patients is needed for each group, 80 patients in total. The comparison will be made using Mann-Whitney U-test.
Who Masked: Participant, Investigator
Masking Description: Both solutions will be kept in identical syringes with an atomization tip (Teflex, MAD Nasal™ Intranasal Mucosal Atomization Device). Each product has a randomized serial number. Both the investigator and the participant are masked. The solutions are made by a different investigator who is not part of the clinical examination, questionnaire filling, patients selection, and recruitment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buffered lidocaine (Experimental): Each participant receives a single intranasal application of atomized 1 mL lidocaine 5% solution combined with bicarbonate 8.4% in a 1:10 ratio.
  Interventions: Drug: Lidocain
- Plain lidocaine (Experimental): Each participant receives a single intranasal application of atomized 1 mL lidocaine 5% solution.
  Interventions: Drug: Lidocain

INTERVENTIONS:
Drug: Lidocain — Layngeal direct fiberoptic examination transnasaly
  Other Names: Transnasal fiberoptic larnyngoscopy

SUMMARY:
Transnasal Fiberoptic Laryngoscopy (TFL) is a common procedure in the otolaryngology clinic for the examination of vocal cord appearance and function, inspection and follow up of benign and malignant lesions, and investigating foreign body ingestion.

There are many forms for applying preprocedural local nasal anesthesia such as atomizers, nebulizers, spray, soaked pads, or local anesthetic gel application.

This study compares the effect of buffered versus plain lidocaine for local nasal anesthesia.

DETAILED DESCRIPTION:
Transnasal Fiberoptic Laryngoscopy (TFL) is a common procedure in the otolaryngology clinic for the examination of vocal cord appearance and function, inspection and follow up of benign and malignant lesions, and investigating foreign body ingestion.

There are many forms for applying preprocedural local nasal anesthesia such as atomizers, nebulizers, spray, soaked pads, or local anesthetic gel application.

Products containing lidocaine are used in everyday practice, sometimes combined with vasoconstrictors such as oxymetazoline or phenylephrine. Lidocaine does not require special storage conditions and is a relatively inexpensive product.

Besides its use for local nasal anesthesia, lidocaine is also widely used for local and regional anesthesia in dentistry, emergency medicine, and surgical or invasive procedures. The addition of bicarbonate for lowering the acidity level of the solution has been studied before in these applications. The buffered solution demonstrated decreased patients pain and increased patient preference[1,2].

Solutions containing lidocaine with a vasoconstrictor such as epinephrine are widely used for soft tissue injection. This combination allows the benefits of prolonged anesthetic and decreased bleeding of the surgical site. However, this combination disadvantage includes increased acidity of the solutions, which may cause increased pain or burning sensation during drug administration. Alkalinization of combined lidocaine and epinephrine solutions has shown decreased local site pain, shorter onset time, and longer duration of anesthesia[3]. The addition of bicarbonate may be done by mixing into a syringe or other suitable container in a relatively easy and fast application for clinical use. Alternatively, a designated device may be used, such as the Onpharma mixing system (Onpharma), commonly used in dentistry[4].

While the alkalinization of lidocaine had shown advantages in local injection into soft tissues, its efficacy for local nasal anesthesia was not previously examined.

This study compares the effect of buffered versus plain lidocaine for local nasal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TFL exam as part of their medical investigation and treatment.
* Age above 18 years and under 65 years.
* Both sexes

Exclusion Criteria:

* Age under 18 years or above 65 years.
* Hypersensitivity to the experiment drugs- bicarbonate, lidocaine, or another drug from the Amid type local anesthetics group (such as Emla or bupivacaine).
* Pregnancy or lactation.
* Signs and symptoms of recent URTI (rhinitis, cough, fever, sinusitis, tonsillitis, pharyngitis).
* Recurrent epistaxis - once per year or more.
* Cardiovascular conditions- ischemic heart disease with decreased physical functions of climbing two staircases or walking 500 meters on a horizontal plane without difficulty. Arrhythmias including permanent or paroxysmal atrial fibrillation, or using a pacemaker.
* Dysphagia- difficulty with swallowing, recurrent aspirations or pneumonia, decreased sensation that may affect swallowing such as previous CVA, peripheral neuropathy from any reason including diabetes. Partial or complete vocal cord immobility.
* Previous TFL exam once in the past six months or twice in the past year.
* Anxiety disorder - with or without drug therapy.
* Recurrent syncope for any reason, including vasovagal syncope. Epilepsy or recurrent seizures.
* Nose and sinuses disease- chronic sinusitis, recurrent sinusitis four or more events per year, Surgical intervention of nose or sinuses in the past year including submucous resection of the septum, turbinectomy, or endoscopic sinus surgery.
* Daily use of a nasal spray of any kind- including steroids or vasoconstrictors.
* Oncologic patients- undergoing chemotherapy or radiation, known tumor in the present or past of the nose and sinuses, nasopharynx, pharynx, hypopharynx, larynx, or subglottis. Patients after resections in these areas or after radiation to head, neck, or chest.
* Severe kidney impairment- GFR under 30 mL/min or severe liver impairment.
* Systemic disease involving the upper airways (e.g. pemphigus).
* Immunosuppression- HIV, drug-induced or congenital
* Unable to give informed consent for any reason, including unable to read or understand the consent form, being under psychiatric assessment, or taking psychiatric drugs.
* Current therapy with known interaction to the experimental drugs- cimetidine, propranolol, phenytoin.
* Moderate to severe nasal polyposis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
VAS- Visual Analogue Scale | Immediately after the procedure
  pain assessment from TFL on a 0-100 visual scale
First symptoms questionnaire | Immediately after the procedure
  pain or burning sensation from local anesthetic administration, bitter or unpleasant taste, suffocation or foreign body sensation of throat, dyspnea, cough, difficulty swallowing saliva, nausea, headache, numbness of mouth and lips, general discomfort during the procedure, patient willingness to go through the procedure again if medically relevant, patient willingness to recommend this procedure to another person if medically relevant. All answers are filled on a 0 to 10 scale, with ten being the most severe.
Second symptoms questionnaire | one hour after TFL exam
  suffocation or foreign body sensation of throat, dyspnea, cough, difficulty swallowing saliva, nausea, headache, numbness of mouth and lips, general discomfort during the procedure, patient willingness to go through the procedure again if medically relevant, patient willingness to recommend this procedure to another person if medically relevant. All answers are filled on a 0 to 10 scale, with ten being the most severe. Duration until symptoms had passed 0-15, 15-30, 30-45, 45-60, 60 minutes or more.
Third questionnaire | one month
  The third questionnaire is filled during a follow-up telephone interview. The patient is asked if there was any epistaxis, syncope, or any other adverse event during the one-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Kfir Kfir, MD, Principal Investigator — Emek Medical Center, Afula, Israel.
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cepeda MS, Tzortzopoulou A, Thackrey M, Hudcova J, Arora Gandhi P, Schumann R. Adjusting the pH of lidocaine for reducing pain on injection. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD006581. doi: 10.1002/14651858.CD006581.pub2. PMID 21154371
- [Background] Lee HJ, Cho YJ, Gong HS, Rhee SH, Park HS, Baek GH. The effect of buffered lidocaine in local anesthesia: a prospective, randomized, double-blind study. J Hand Surg Am. 2013 May;38(5):971-5. doi: 10.1016/j.jhsa.2013.02.016. Epub 2013 Apr 6. PMID 23566722
- [Background] Gupta S, Kumar A, Sharma AK, Purohit J, Narula JS. "Sodium bicarbonate": an adjunct to painless palatal anesthesia. Oral Maxillofac Surg. 2018 Dec;22(4):451-455. doi: 10.1007/s10006-018-0730-x. Epub 2018 Oct 15. PMID 30324508
- [Background] Goodchild JH, Donaldson M. Novel Direct Injection Chairside Buffering Technique for Local Anesthetic Use in Dentistry. Compend Contin Educ Dent. 2019 Jul/Aug;40(7):e1-e10. PMID 31478693
- [Background] Nakayama M, Munemura Y, Kanaya N, Tsuchida H, Namiki A. Efficacy of alkalinized lidocaine for reducing pain on intravenous and epidural catheterization. J Anesth. 2001;15(4):201-3. doi: 10.1007/s005400170003. PMID 14569436